CLINICAL TRIAL: NCT04020744
Title: Targeting Hippocampal Hyperactivity With Real-time Functional MRI Based Neurofeedback in Elderly Individuals With and Without Memory Problems
Brief Title: Real-time fMRI Neurofeedback in Patients With MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1163
Record Dates: First submitted 2019-07-04; First posted 2019-07-16 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Masking Description: For blinding of the participants, they will be told that they will be asked to regulate one of two brain regions, without mentioning the specific area.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- healthy elderly participants receiving feedback from the hippocampus (Active Comparator): This group will consist of healthy elderly volunteers, who will receive feedback from their hippocampal activity.
  Interventions: Other: real-time fMRI based neurofeedback from the hippocampus
- healthy elderly participants receiving feedback from another area (Sham Comparator): This group will consist of healthy elderly volunteers, who will receive feedback from another brain area.
  Interventions: Other: real-time fMRI based neurofeedback from another brain area
- patients with MCI receiving feedback from the hippocampus (Experimental): This group will consist of patients with mild cognitive impairment, who will receive feedback from their hippocampal activity.
  Interventions: Other: real-time fMRI based neurofeedback from the hippocampus
- patients with MCI receiving feedback from another brain area (Sham Comparator): This group will consist of patients with mild cognitive impairment, who will receive feedback from another brain area.
  Interventions: Other: real-time fMRI based neurofeedback from another brain area

INTERVENTIONS:
Other: real-time fMRI based neurofeedback from the hippocampus — During real-time fMRI neurofeedback, participants are trained to 'control' hippocampal activity. The training is accomplished by continuously measuring brain activity, analysing it in real-time, and then providing feedback about the current (and the targeted) brain activity to the participant.
  Arms: healthy elderly participants receiving feedback from the hippocampus; patients with MCI receiving feedback from the hippocampus
Other: real-time fMRI based neurofeedback from another brain area — During real-time fMRI neurofeedback, participants are trained to 'control' hippocampal activity. The training is accomplished by continuously measuring brain activity, analysing it in real-time, and then providing feedback about the current (and the targeted) brain activity to the participant.
  Arms: healthy elderly participants receiving feedback from another area; patients with MCI receiving feedback from another brain area

SUMMARY:
Increased activity in the hippocampus (i.e., hyperactivity) during a fMRI memory task was found in patients with Mild Cognitive Impairment due to Alzheimer's disease (MCI). Those with increased hippocampal activity exhibited elevated clinical progression. Reducing hippocampal hyperactivity with pharmacological treatment reduced hyperactivity and improved memory performance. The investigators of this study will test whether real-time fMRI neurofeedback will also downregulate hippocampal activity and thereby improve memory performance.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is an insidious and progressive neurodegenerative disorder accompanied by extracellular deposits of beta-amyloid ( aβ) and the increase of cognitive dysfunctions. Several functional magnet resonance imaging (fMRI) studies in the prodromal stage of AD (i.e., in MCI) have found increased hippocampal activity during a memory task to be predictive of memory worsening and disease progression. In this study the investigators are aiming to reduce hippocampal hyperactivity with real-time fMRI neurofeedback and test whether this will improve memory performance.

This study will use a randomized, single-blind, parallel group design. Patients with MCI and healthy participants will be assigned to receive feedback from either the hippocampus (experimental group, N=42) or from another brain area (alternate ROI feedback group, N=42). All participants will be instructed to downregulate activity.

ELIGIBILITY:
Inclusion Criteria:

* Intact activities of daily living
* Fluent in German
* Normal/corrected-to-normal vision
* Written informed consent

Exclusion Criteria:

* Dementia
* Current/lifetime severe psychiatric or neurological disorder
* History of seizures
* Psychotropic medication
* Currently/lifetime drug or alcohol abuse
* Brain damage
* Magnetisable implants

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Rate of change in hippocampal activity during a memory task | Directly after the intervention
  Measured by fMRI (rate of change in activity from baseline to after the intervention)

SECONDARY OUTCOMES:
Rate of change in memory performance | Directly after the intervention
  Measured by fMRI (memory performance change from baseline to after the intervention)
Rate of change from in memory performance (behavioural) | Directly after the intervention
  Measured behaviourally (memory performance change from baseline to after the intervention)

OTHER OUTCOMES:
Strategies for Regulation of hippocampal activity | Intervention
  Which strategies were particularly helpful in downregulation of hippocampal activity (number of times the strategies were mentioned)
Predictors of neurofeedback success | Post-Intervention
  Variables extracted from questionnaires that may predict who will respond to neurofeedback

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Peter, PD Dr., Principal Investigator — University of Bern; Stefan Klöppel, Prof. Dr., Principal Investigator — University of Bern; Frank Scharnowski, Prof. Dr., Study Chair — University of Vienna; Roland Wiest, Prof. Dr., Study Chair — University of Bern; Katharina Klink, Study Chair — University of Bern
Locations (2):
- Switzerland (2):
  - SITEM (Swiss Institute for Translational and Entrepreneurial Medicine), Bern
  - University of Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klink K, Jaun U, Federspiel A, Wunderlin M, Teunissen CE, Kiefer C, Wiest R, Scharnowski F, Sladky R, Haugg A, Hellrung L, Peter J. Targeting hippocampal hyperactivity with real-time fMRI neurofeedback: protocol of a single-blind randomized controlled trial in mild cognitive impairment. BMC Psychiatry. 2021 Feb 9;21(1):87. doi: 10.1186/s12888-021-03091-8. PMID 33563242